CLINICAL TRIAL: NCT02290821
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Diclofenac Sodium Topical Gel (DSG) 1% Applied Four Times Daily in Subjects With Acute Blunt Soft Tissue Injuries/Contusions of the Limbs
Brief Title: Efficacy and Safety of Diclofenac Sodium Topical Gel 1% Compared to Placebo in Subjects With Acute Blunt Trauma Injuries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 197-P-322
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: Acute Blunt Soft Tissue Injuries/Contusions
MeSH Terms: conditions — Contusions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac sodium gel 1% (Experimental): diclofenac sodium gel 1%
  Interventions: Drug: placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: placebo
  Arms: diclofenac sodium gel 1%
Drug: Placebos
  Arms: Placebo

SUMMARY:
This study will assess the analgesic efficacy of DSG 1% compared to placebo in the reduction of the pain associated with acute blunt trauma injuries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 16 years and over Fresh impact injury of the upper or lower limbs, not requiring admittance to hospital & meeting baseline pain intensity level Anticipated time between injury and treatment must be ≤ 6 hours

Exclusion Criteria:

* Pain medication prior to randomization Topical analgesic or anti-inflammatory treatment over the previous month in the area to be treated Any physical impairment that would influence efficacy assessments, such as peripheral or central neurological disease, significant back pain, painful conditions of the upper or lower extremities Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - US Site, Bradenton, Florida
  - US Site, Port Orange, Florida
  - US Site, Boise, Idaho
  - US Site, Grand Rapids, Michigan
  - US Site, Omaha, Nebraska
  - US Site, Brooklyn, New York
  - US Site, Columbus, Ohio
  - US Site, State College, Pennsylvania
  - US Site, Bellaine, Texas
  - US Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  diclofenac sodium gel 1%
Period: Overall Study
Arm/Group | Diclofenac Sodium Gel 1% | Placebo
Started | 109 | 106
Completed | 103 | 103
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Unable or unwilling to cooperate with | 2 | 0
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Gel 1% | Placebo | Total
Number analyzed (Participants) | 109 | 106 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (10.7) | 26.3 (8.5) | 26.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 92 | 82 | 174
Region of Enrollment [Number; unit: participants]
  United States | 109 | 106 | 215

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Differences Over 24 Hours After Initiating Treatment (SPID 24)
Description: The primary efficacy outcome was the time-weighted SPID 24 (POW). Sum of pain intensity differences over 24 hours after initiating treatment (SPID 24) for the ITT population. SPID 24 derived from spontaneous Pain Intensity scores assessed over 24 hours on a 0 (No pain) - 10 (Pain as bad as you can imagine) Numerical Rating Scale. SPID 24 was computed using the trapezoidal rule, i.e. Σ [T(i) - T(i-1)] x [((PID)(i-1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time i, is the baseline pain intensity (PI) score - PI score at Time i. Scores were assessed hourly for the first 4 hours and then every 2 hours whilst subjects were awake. Linear interpolation was used to compute an exact SPID as of 24 hours. SPID-24 was computed after all imputation of missing assessments and post-rescue assessments had been completed.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diclofenac Sodium Gel 1% | Placebo
Number analyzed (Participants) | 109 | 106
units on a scale | 42.9 (40.6) | 45.5 (42.6)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Diclofenac Sodium Gel 1% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/106
Other Adverse Events (participants affected / at risk) | 4/109 | 2/106
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Gel 1% (N=109) | Placebo (N=106)
headache (Nervous system disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator